CLINICAL TRIAL: NCT03897621
Title: The Effect of Tranexamic Acid on Blood Coagulation in Total Hip Arthroplasty Surgery Based on Rotational Thromboelastometry (ROTEM®).
Brief Title: The Effect of Tranexamic Acid on Blood Coagulation in Total Hip Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Uzung Yoon, Clinical Instructor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18D.581
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Coagulation; Intravascular; Rotational Thromboelastometry; Fibrinolysis; Hemorrhage; Tranexamic Acid; Total Hip Arthroplasty
Keywords: tranexamic acid; Rotational thromboelastometry; Fibrinolysis; viscoelastic essay
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: double-blinded randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid (Experimental): Patients undergoing unilateral, primary, total hip arthroplasty with English as their native language
  Interventions: Drug: Tranexamic Acid
- Normal saline (Placebo Comparator): Patients undergoing unilateral, primary, total hip arthroplasty with English as their native language
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — tranexamic acid will be administered intravenously after induction of anesthesia (a bolus of 10 mg/kg or maximal dose of 1g).
  Arms: tranexamic acid
Drug: Placebo — Patients in the placebo group will receive normal saline (a bolus of sodium chloride 0.9%, 0.1 mL/kg or maximal dose of 10 mL).
  Arms: Normal saline

SUMMARY:
Total hip arthroplasty (THA) is associated with blood loss ranging from 300 to 2000 mL. Tranexamic acid (TXA) is frequently administered prophylactically during this procedure to reduce blood loss by inhibiting fibrinolysis or by stopping naturally occurring clot resolution. TXA is employed currently based on a surgeon's preference. The objective of this study is to quantitate the degree of fibrinolysis using rotational thromboelastometry (ROTEM) and investigate the role of TXA prophylaxis on blood loss in patients undergoing THA in a double-blind fashion. Our hypothesis is that fibrinolysis is minimal at most and TXA prophylaxis is not necessary during THA. All patients, whether they receive TXA or normal saline, will not be at risk, as at this time no data exists to determine which approach is safer or more effective. This is the first study to compare TXA vs. placebo in a double-blinded, randomized controlled trial.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is associated with moderate blood loss ranging from 300 to 2000 mL. Tranexamic acid (TXA) is frequently administered prophylactically during this procedure to reduce blood loss by inhibiting fibrinolysis. Most clinical studies reported potential benefit of the treatment demonstrated by less estimated blood loss (EBL), reduced hemoglobin/hematocrit (HH) change, and reduced transfused packed red blood cells (PRBC). However, bleeding complication may be affected more significantly by the degree of surgical trauma and comorbidity of patients than coagulation abnormality. Further, the frequency and severity of fibrinolysis during these procedures have not been well studied. Additionally, TXA administration may increase the tendency of postoperative venous thrombosis by inhibiting fibrinolysis in already prothrombotic patients. The objective of this study is to quantitate the degree of fibrinolysis using rotational thromboelastometry (ROTEM) and investigate the role of TXA prophylaxis on clinical outcome in patients undergoing THA in a double-blind fashion. Our hypothesis is that fibrinolysis is minimal at most and TXA prophylaxis is not necessary during primary THA.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include total of 200 adults (age range of 18 - 85 years) who are in the American Society of Anesthesiologists (ASA) Physical Status (PS) 1-3. Inclusion criteria are patients undergoing unilateral, primary, total hip arthroplasty.

Exclusion Criteria:

* Exclusion criteria include patient's refusal, patients with history of significant coagulopathy or on anticoagulation therapy. Female patients who are pregnant or nursing will be excluded. In addition, patients with anemia (Hb < 8 g/dL) or who received blood transfusion within one week before surgery will be excluded. Patient receiving subcutaneous heparin on the same day prior to surgery will be also excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Fibrinolysis | after induction of anesthesia (baseline),
  Fibrinolysis based on ROTEM parameter, defined as ML (maxium lysis) >15%
Fibrinolysis | 45 min after drug administration,
  Fibrinolysis based on ROTEM parameter, defined as ML (maxium lysis) >15%
Fibrinolysis | one hour after the end of surgery
  Fibrinolysis based on ROTEM parameter, defined as ML (maxium lysis) >15%

SECONDARY OUTCOMES:
Blood loss | during surgery (intraoperative)
  amount of blood loss in milliliter during surgery
blood transfusion | Intraoperative and up to 72-hour after surgery
  Amount of Packed Red Blood Cells (PRBC) transfused
pre- and postoperative hemoglobin level | up to 72-hour after surgery
  Pre and postoperative hemoglobin level in grams per deciliter
Wound infection | up to 72-hour after surgery
  Incidence of wound infection
Hematoma | up to72-hour after surgery
  Incidence of hematoma
Thrombotic events (PE, DVT). | up to 72-hour after surgery
  Incidence of thrombotic events (pulmonary embolism, deep vein thrombosis)

CONTACTS AND LOCATIONS:
Overall Officials: Uzung Yoon, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu Y, Yang T, Zeng Y, Si H, Cao F, Shen B. Tranexamic acid reduces blood loss and transfusion requirements in primary simultaneous bilateral total knee arthroplasty: a meta-analysis of randomized controlled trials. Blood Coagul Fibrinolysis. 2017 Oct;28(7):501-508. doi: 10.1097/MBC.0000000000000637. PMID 28448319
- [Result] Prieto HA, Vincent HK, Deen JT, Iams DA, Parvataneni HK. Tranexamic Acid Effectively Reduces Blood Loss and Transfusion Rates during Simultaneous Bilateral Total Knee Arthroplasty. J Knee Surg. 2018 Mar;31(3):270-276. doi: 10.1055/s-0037-1603333. Epub 2017 May 15. PMID 28505683
- [Result] Na HS, Shin HJ, Lee YJ, Kim JH, Koo KH, Do SH. The effect of tranexamic acid on blood coagulation in total hip replacement arthroplasty: rotational thromboelastographic (ROTEM(R)) analysis. Anaesthesia. 2016 Jan;71(1):67-75. doi: 10.1111/anae.13270. Epub 2015 Nov 12. PMID 26559015
- [Result] Watts CD, Houdek MT, Sems SA, Cross WW, Pagnano MW. Tranexamic Acid Safely Reduced Blood Loss in Hemi- and Total Hip Arthroplasty for Acute Femoral Neck Fracture: A Randomized Clinical Trial. J Orthop Trauma. 2017 Jul;31(7):345-351. doi: 10.1097/BOT.0000000000000837. PMID 28633147
- [Result] Zufferey PJ, Lanoiselee J, Chapelle C, Borisov DB, Bien JY, Lambert P, Philippot R, Molliex S, Delavenne X; investigators of the PeriOpeRative Tranexamic acid in hip arthrOplasty (PORTO) Study. Intravenous Tranexamic Acid Bolus plus Infusion Is Not More Effective than a Single Bolus in Primary Hip Arthroplasty: A Randomized Controlled Trial. Anesthesiology. 2017 Sep;127(3):413-422. doi: 10.1097/ALN.0000000000001787. PMID 28692467
- [Result] Toledo P, McCarthy RJ, Hewlett BJ, Fitzgerald PC, Wong CA. The accuracy of blood loss estimation after simulated vaginal delivery. Anesth Analg. 2007 Dec;105(6):1736-40, table of contents. doi: 10.1213/01.ane.0000286233.48111.d8. PMID 18042876
- [Result] Brecher ME, Monk T, Goodnough LT. A standardized method for calculating blood loss. Transfusion. 1997 Oct;37(10):1070-4. doi: 10.1046/j.1537-2995.1997.371098016448.x. PMID 9354828
- [Result] Theusinger OM, Wanner GA, Emmert MY, Billeter A, Eismon J, Seifert B, Simmen HP, Spahn DR, Baulig W. Hyperfibrinolysis diagnosed by rotational thromboelastometry (ROTEM) is associated with higher mortality in patients with severe trauma. Anesth Analg. 2011 Nov;113(5):1003-12. doi: 10.1213/ANE.0b013e31822e183f. Epub 2011 Sep 14. PMID 21918164
- [Result] Ram GG, Suresh P, Vijayaraghavan PV. Surgeons often underestimate the amount of blood loss in replacement surgeries. Chin J Traumatol. 2014;17(4):225-8. PMID 25098850
- [Result] Levrat A, Gros A, Rugeri L, Inaba K, Floccard B, Negrier C, David JS. Evaluation of rotation thrombelastography for the diagnosis of hyperfibrinolysis in trauma patients. Br J Anaesth. 2008 Jun;100(6):792-7. doi: 10.1093/bja/aen083. Epub 2008 Apr 24. PMID 18440953
- [Derived] Yoon U, Beausang D, Elia E, Torjman M, Mojica J, Purtill J, Nazarian D, Courtney PM, Kang Y. The effect of tranexamic acid on blood coagulation in primary total hip arthroplasty using rotational thromboelastometry: a randomized controlled trial. EClinicalMedicine. 2025 Jul 21;86:103374. doi: 10.1016/j.eclinm.2025.103374. eCollection 2025 Aug. PMID 40735345